CLINICAL TRIAL: NCT02515162
Title: Fischer Cone Biopsy Excisor Versus Loop Excision Procedure. A Randomized Trial of Two Operation Techniques in Women Undergoing Conization for Cervical Dysplasia
Brief Title: Fischer Cone Biopsy Excisor Versus Loop Excision Procedure for Conization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Collaborators: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Dr. med. Ziad Hilal, Dr. med. Ziad Hilal, Zydolab - Institute of Cytology and Immune Cytochemistry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONE-2
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Uterine Cervical Dysplasia
Keywords: conization; LLETZ; cervical dysplasia; cervical intraepithelial neoplasia; Fischer cone biopsy excisor; loop electrosurgical excision procedure
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fischer Cone Biopsy Excisor (Experimental): Conization Methode using a triangular electrode , i.e. Fischer Cone Biopsy Excisor
  Interventions: Procedure: Fischer Cone Biopsy Excisor
- Loop Excision Procedure (Active Comparator): Conization Methode using a circular electrode , i.e. Loop excision Procedure
  Interventions: Procedure: Loop Excision Procedure

INTERVENTIONS:
Procedure: Fischer Cone Biopsy Excisor — Electrosurgical excision method using a triangular electrode to remove the abnormal cervical Transformation zone
  Arms: Fischer Cone Biopsy Excisor
Procedure: Loop Excision Procedure — Electrosurgical excision method using a circular electrode to remove the abnormal cervical Transformation zone
  Arms: Loop Excision Procedure

SUMMARY:
In a randomized clinical trial of 160 women undergoing conization for cervical dysplasia, two electrosurgical excision methods, Fischer Cone Biopsy Excison vs. Loop Excision Procedure, will be compared. The primary outcome of the study is dysplasia-free resection margin rate, secondary outcomes are intraoperative blood loss, time to complete hemostasis, intervention time, postoperative pain, intra- and postoperative complications, the resected cone volume and users satisfaction.

DETAILED DESCRIPTION:
Conization is the method of choice in therapy for cervical dysplasia. Beside the risk of preterm delivery, the risk of a local relapse in patients with dysplasia-affected resection margin is high.

The Goldstandard standard technique in conization for women with cervical dysplasia is the large loop excision of the transformation zone ("LLETZ"). Nevertheless other techniques such as the excision of the abnormal tissue with the so called "Fischer Cone Biopsy Excisor" could provide advantages and is yet not enough investigated. The loop excision technique uses a circular electrode, in contrast Fischer Cone Biopsy Excision is done by a triangular electrode.

It is unknown, whether the use of the circular or the triangular electrode is superior regarding the dysplasia-free resection margin rate and other outcome parameters such as the resected cone volume, postoperative bleeding and postoperative pain. Therefore, the investigator designed a randomized clinical trial of 160 women undergoing conization for cervical dysplasia, comparing the two electrosurgical techniques, "LLETZ-conization" and "Fischer Cone Biopsy Excision". The primary outcome of the study is the dysplasia-free resection margin rate independently proved by a pathologist, secondary outcomes are intraoperative blood loss measured as difference in serum hemoglobin pre- and postoperatively, postoperative pain according to a 11 step VAS scale, time to complete hemostasis measured in seconds, duration of the intervention measured in minutes, resected cone volume, users satisfaction according to a 11 step VAS scale and intra- and postoperative complications, defined as necessity to intervene surgically up to 14 days postoperatively.

The study Population consists of women undergoing conization for histologically proven cervical dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven cervical dysplasia
* colposcopy Prior to conization
* informed consent
* no known hematologic disorder

Exclusion Criteria:

* significant language barrier
* a personal history of conization
* pregnancy
* the use of blood thinner
* unwillingness to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Margin status | 2 Days after conization
  Resection margin is judge as "R0" if abnormal cells are not found in the margin of the biopsy or "R1" if abnormal cells remain in the margin of the biopsy. The histopathological examination will be done by an Independent pathologist

SECONDARY OUTCOMES:
Intraoperative blood loss | 5 hours
  intraoperative blood loss will be measured using the difference in serum hemoglobin one day prior to surgery and within 5 hours postoperatively
Postoperative pain | 5 hours
  patients will score their postoperative pain Level using a 11-step visual analogue scale (nVAS) and a 5-step graphical visual analogue scale (gVAS)within 5 hours after surgery
Time to complete intraoperative hemostasis | 120 seconds
  the time until complete hemostasis as judged by the surgeon has been achieved, will be measured in seconds
Operation time | 20 minutes
  the time from the beginning of the Operation (start of the electrosurgical method) until the end of the operation (the end of hemostatic interventions) will be measured in minutes
Resected cone volume | 10 minutes
  The resected cone volume will be measured postoperative by using a scale
satisfaction with the device | 30 minutes
  surgeons will score their preference regarding the surgical method using an 11-step visual analogue scale (VAS) for ,satisfaction with the device' (ranging from 0 (,very satisfied') to 10 (,absolutely not satisfied')
handling of the device | 30 minutes
  surgeons will score their preference regarding the surgical method using an 11-step visual analogue scale (VAS) for ,(ranging from 0 (,very easy') to 10 (,very difficult')
Operative complications | 14 days
  Operative complications defined as necessity to intervene surgically up to 14 days postoperatively
number of fragments of the surgical specimen | 10 minutes
  surgeons will count the number of the surgical specimen (1 vs. >1)

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hilal, Dr. med., Principal Investigator — Zydolab - Institute of Cytology and Immune Cytochemistry
Locations (1):
- Department of Obstetrics and Gynecology of the Ruhr University Bochum, Herne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bevis KS, Biggio JR. Cervical conization and the risk of preterm delivery. Am J Obstet Gynecol. 2011 Jul;205(1):19-27. doi: 10.1016/j.ajog.2011.01.003. Epub 2011 Feb 23. PMID 21345402
- [Background] Jin G, LanLan Z, Li C, Dan Z. Pregnancy outcome following loop electrosurgical excision procedure (LEEP) a systematic review and meta-analysis. Arch Gynecol Obstet. 2014 Jan;289(1):85-99. doi: 10.1007/s00404-013-2955-0. Epub 2013 Jul 11. PMID 23843155
- [Background] Khalid S, Dimitriou E, Conroy R, Paraskevaidis E, Kyrgiou M, Harrity C, Arbyn M, Prendiville W. The thickness and volume of LLETZ specimens can predict the relative risk of pregnancy-related morbidity. BJOG. 2012 May;119(6):685-91. doi: 10.1111/j.1471-0528.2011.03252.x. Epub 2012 Feb 14. PMID 22329499
- [Background] Shaco-Levy R, Eger G, Dreiher J, Benharroch D, Meirovitz M. Positive margin status in uterine cervix cone specimens is associated with persistent/recurrent high-grade dysplasia. Int J Gynecol Pathol. 2014 Jan;33(1):83-8. doi: 10.1097/PGP.0b013e3182763158. PMID 24300540
- [Background] Mathevet P, Chemali E, Roy M, Dargent D. Long-term outcome of a randomized study comparing three techniques of conization: cold knife, laser, and LEEP. Eur J Obstet Gynecol Reprod Biol. 2003 Feb 10;106(2):214-8. doi: 10.1016/s0301-2115(02)00245-2. PMID 12551795
- [Background] Boardman LA, Steinhoff MM, Shackelton R, Weitzen S, Crowthers L. A randomized trial of the Fischer cone biopsy excisor and loop electrosurgical excision procedure. Obstet Gynecol. 2004 Oct;104(4):745-50. doi: 10.1097/01.AOG.0000139517.26003.fc. PMID 15458896